CLINICAL TRIAL: NCT05567939
Title: Clinical, Virological, Serological and Psychosocial Outcomes in Human Monkeypox Virus Infectious Disease - a PROspective Observational Cohort Study for Epidemiology and Outcomes of MPXVID
Brief Title: Clinical, Virological, Immunological, Psychosocial and Epidemiological Consequences of Human Monkeypox Virus (ProMPX)
Acronym: ProMPX
Status: Terminated | Type: Observational
Why Stopped: Due to the decrease in the number of mpox infections in the Netherlands, we were unable to include the desired number of study participants.
Sponsor: Public Health Service of Amsterdam (Other Government)
Responsible Party: Principal Investigator, Henry J.C. de Vries, Professor Doctor, Public Health Service of Amsterdam
Other Study IDs: ProMPX
Record Dates: First submitted 2022-09-27; First posted 2022-10-05 (Actual); Last update posted 2024-06-03 (Actual); Status verified 2024-05

CONDITIONS: Monkeypox; Monkey Pox
MeSH Terms: conditions — Mpox, Monkeypox

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case: Individuals with laboratory confirmed MPXVID
  Interventions: Other: Natural course of disease
- Control: Individuals without proctitis and without MPXVID-related symptoms
  Interventions: Other: Natural course of disease

INTERVENTIONS:
Other: Natural course of disease — Sample and questionnaire collection

SUMMARY:
MonkeyPox Virus Infectious Disease (MPXVID) is a viral infection caused by the monkeypox virus (MPXV) which is an orthopoxvirus that is endemic in countries in West and Central Africa. The clinical course of the MPXVID is similar to smallpox (variola) but usually milder - with less severe disease symptoms seen in the West African subtype. Historically, the case fatality ratio of MPXVID ranged from 0 to 11% and fatality occurs more commonly among children. In Europe, human MPXVID only occurred as an imported disease with limited onward transmission. However, since May 2022 over 19.000 cases of MPXVID - mostly with the West African subtype - have been reported in Europe without a travel history to the endemic areas in Africa. The far large majority of patients with MPXVID in the current outbreak are gay, bisexual and other men who have sex with men (GBMSM). There is an urgent need to address essential knowledge gaps for optimal clinical care and public health management.

The aim of this study is to improve our understanding of clinical, virological, and psychosocial outcomes in patients with MPXVID. To get a better understanding of associated risk factors for MPXV infection, and to measure quality of life and stigma, the investigators will also include a control population of men without proctitis and MPXVID-related symptoms at day 0. In addition, the investigators want to assess the vaccine effectiveness against MPXVID of infant smallpox vaccination given before 1974, as well as vaccine effectiveness of the modified vaccinia Ankara (MVA) smallpox vaccine, when administered as pre- or post-exposure prophylaxis in high risk contacts of MPXVD patients.

ELIGIBILITY:
Inclusion Criteria

Case:

- Individuals, with: I. Laboratory confirmed MPXVID, or II. A presumptive MPXVID case with pending laboratory confirmation

- Be able to provide informed consent by means of: I. Verbal or deferred informed consent, which will be complemented with a written informed consent during the subsequent outpatient study visit; II. Written informed consent during the baseline visit for presumptive cases

- Sufficient understanding of the Dutch or English language.

Control:

- Individuals without proctitis and MPXVID-related symptoms

Exclusion Criteria

Case:

* Presumptive cases with subsequent negative test for MPXV (can be included as control);
* Being under the age of 16 years old;
* Unlikely to comply with the study procedures, as deemed by the recruiting research doctor/nurse;
* Mental disorder that in the view of the investigator would interfere with adherence to the study procedures, or the decision to participate in the study;
* Investigators or otherwise dependent persons;
* Living in long term care facility.

Control:

* Positive test result for MPXV at baseline (day 0)
* Being under the age of 16 years old;
* Unlikely to comply with the study procedures, as deemed by the recruiting research doctor/nurse;
* Mental disorder that in the view of the investigator would interfere with adherence to the study procedures, or the decision to participate in the study;
* Investigators or otherwise dependent persons;
* Living in long term care facility.

Min Age: 16 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: The target population are all individuals visiting the STI-clinic of the Public Health Services of Amsterdam, irrespective of their gender, aged 16 years or older with a laboratory confirmed MPXV infection, or are suspected of MPXV while laboratory confirmation is pending. MPXV infection is diagnosed according to a routinely performed PCR test on lesion, anal-, pharyngeal and vaginal swabs in patients suspect of having MPXVID. The controls will be clients of the STI clinic who are individuals without proctitis and without MPXVID-related symptoms; they will only be matched on date of inclusion.
Sampling Method: Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2022-09-19 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
What is the time to resolution of symptoms among patients with symptomatic MPXVID? | 28 days
  The time between appearance of the first lesions and the day on which all skin lesions are epithelialized and crusts fall off, and all systemic symptoms (incl. proctitis) have resolved.

SECONDARY OUTCOMES:
To describe and analyse demographic characteristics in patients with MPXVID. | 180 days
  Demographic characteristics at enrolment visit.
To describe and analyse sexual characteristics in patients with MPXVID. | 180 days
  Sexual characteristics at enrolment visit.
To describe and analyse clinical characteristics in patients with MPXVID. | 180 days
  Clinical status of MPXVID at baseline and days 4, 8, 14, 21, 60 and 180:
  * According to a 4 pt ordinal scale.
  * Location(s) of lesion(s): peri-genital, peri-anal, peri-oral, romp, arms, legs, head.
  * Number of lesions: 1, 2-5, >5.
  * Presence of proctitis related symptoms.
To describe and analyse other clinical characteristics in patients with MPXVID. | 180 days
  Other clinical outcomes on days 4, 8, 14, 21, 60 and 180, as follows:
  * Proportion of patients with systemic symptoms.
  * Proportion of patients with proctitis.
  * Proportion of patients with oral lesions, pharyngitis and/or oesophagitis
  * Proportion of patients requiring pain medication.
  * Proportion of patients requiring additional medical consultations
  * Proportion of patients with a significant reduction of their quality of live (measured with Dermatology Life Quality Index (DLQI) with outcome above 10 points).
  * Proportion of patients with secondary bacterial infection of MPXVID lesions.
To describe the presence of MPXV DNA and cycle threshold (Ct) values in patients with MPXVID. | 180 days
  The presence of MPXV DNA and cycle threshold (Ct) values in lesion swabs on baseline and days 4, 8, 14, 21 and 28.
To describe other virological outcomes in patients with MPXVID. | 180 days
  Change from baseline in MPXV DNA levels in anal-, pharyngeal and vaginal swabs, semen and blood (also the development of antibody levels) on days 4, 8, 14, 21, 28, 60 and 180.
To describe changes in sexual behaviour in patients with MPXVID in comparison to controls. | 180 days
  Sexual behaviour measurement at baseline and change at days 14, 28, 60 and 180 (only baseline, day 60 and day 180 for controls).
To describe changes in quality of life in patients with MPXVID in comparison to controls. | 180 days
  DLQI questionnaire measurement of the quality of live change at baseline and change at days 14, 28, 60 and 180 (only baseline, day 60 and day 180 for controls).
To describe changes in the experience of (internalized) stigma in patients with MPXVID in comparison to controls. | 180 days
  Questionnaires of the experience of (internalized) stigma at baseline and change at days 28 and 180 (only baseline and day 180 for controls).
To describe changes in the experience of fatigue in patients with MPXVID in comparison to controls. | 60 days
  Sexual Function Questionnaire (SFQ) questionnaire measurement of fatigue at baseline and change at days 14, 28, and 60 (only baseline and day 60 for controls).
To describe changes in the physical and psychological health in patients with MPXVID in comparison to controls. | 180 days
  PATIENT HEALTH QUESTIONNAIRE - Schedule for Affective Disorders and Schizophrenia (PHQ-SADS) questionnaire measurement of anxiety, depression, somatic complaints at baseline and change at days 28 and 180 (only baseline and day 180 for controls).
To estimate the effectiveness against MPXVID of infant smallpox vaccine given before 1974. | through study completion, an average of 1 year
  Measuring the proportion of patients with a laboratory confirmed MPXVID and of controls without MPXVID who are vaccinated with the infant smallpox vaccine before 1974, and estimate vaccine effectiveness (i.e. disease severity outcome).
To estimate the effectiveness against MPXVID of modified vaccinia Ankara (MVA) smallpox vaccine. | through study completion, an average of 1 year
  Measuring the proportion of patients with a laboratory confirmed MPXVID and of controls without MPXVID who are vaccinated with the modified vaccinia Ankara (MVA) smallpox vaccine, either as pre- or as post-exposure prophylaxis against MPX after June 2022.
To describe the use of antiviral medication and/or immunoglobulins. | 180 days
  Proportion of patients treated with antiviral and/or immunoglobulins.

CONTACTS AND LOCATIONS:
Locations (1):
- Public Health Service, Amsterdam, North Holland, Netherlands